CLINICAL TRIAL: NCT06256029
Title: The Effect of Recruitment Maneuver on Static Compliance in Patients Undergoing General Anesthesia for Laparoscopic Cholecystectomy
Brief Title: Recruitment Maneuver in General Anesthesia for Laparoscopic Cholecystectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Novi Sad (Other)
Responsible Party: Principal Investigator, Mihaela Preveden, Principal investigator, University of Novi Sad
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00-39/2023
Record Dates: First submitted 2024-02-04; First posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Mechanical Ventilation Pressure High

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): All participants will undergo the recruitment maneuver. The patients will be divided into non-obese patients (BMI 18.5-24.9 kg/m²) and patients with increased body mass (BMI 25-34.9 kg/m²).
  Interventions: Procedure: Recruitment maneuver

INTERVENTIONS:
Procedure: Recruitment maneuver — The recruitment maneuver will be performed by increasing the current peak pressure (Ppeak) by 5 cm H2O, changing the inspiratory/expiratory ratio from 1:2 to 1:1, with PEEP values of 5 and 7 cm H2O. The respiratory rate during the recruitment maneuver will be 10 breaths per minute, and the recruitment maneuver will last 30 seconds (5 breaths). The recruitment maneuver will be performed 3 times: the first time immediately after the formation of the pneumoperitoneum and the positioning of the patient in the reverse Trendelenburg position with a PEEP of 5 cm H2O, the second time with a PEEP of 7 cm H2O, during the duration of the operation. The third recruitment maneuver will be performed with a PEEP of 7 cm H2O at the end of the operative procedure, and immediately before the patient wakes up. After each increase, PEEP will be maintained at higher pressure values with a peak value of 7 cm H2O.

SUMMARY:
This is a prospective non-randomized clinical trial evaluating the effect of the recruitment maneuver on static compliance in patients undergoing general anesthesia for laparoscopic cholecystectomy

DETAILED DESCRIPTION:
The study will be performed in patients who are scheduled for laparoscopic cholecystectomy. They will be divided into two groups. Group I will consist of non-obese patients (Body Mass Index - BMI from 18.5 to 24.9 kg/m²), while group II will consist of patients with increased body mass (pre-obese and obese class I with BMI from 25 to 34.9 kg/m²).

The recruitment maneuver will be performed by increasing the current peak pressure (Ppeak) by 5 cm H2O, changing the inspiratory/expiratory ratio from 1:2 to 1:1, with PEEP values of 5 and 7 cm H2O. The respiratory rate during the recruitment maneuver will be 10 breaths per minute, and the recruitment maneuver will last 30 seconds (5 breaths). In both groups of patients, the recruitment maneuver will be performed 3 times: the first time immediately after the formation of the pneumoperitoneum and the positioning of the patient in the reverse Trendelenburg position with a PEEP of 5 cm H2O, the second time with a PEEP of 7 cm H2O, during the duration of the operation. The third recruitment maneuver will be performed with a PEEP of 7 cm H2O at the end of the operative procedure, and immediately before the patient wakes up. After each increase, PEEP will be maintained at higher pressure values with a peak value of 7 cm H2O.

Parameters of respiratory mechanics and vital parameters will be monitored during multiple stages of the laparoscopic cholecystectomy, as well as after the recruitment maneuver: (T1) after induction of anesthesia, and before the formation of pneumoperitoneum; (T2) after the formation of pneumoperitoneum and positioning of the patient in reverse Trendelenburg position; (T3) after recruitment maneuver with PEEP values of 5 cm H2O; (T4) after recruitment maneuver with PEEP values of 7 cm H2O; (T5) after deflation; (T6) immediately before awakening with recruitment maneuver and PEEP values of 7 cm H2O. All measurements will be made in VCV mode of mechanical ventilation, and recruitment maneuver will be performed in pressure control ventilation (PCV) mode of mechanical lung ventilation.

The parameters of the respiratory system mechanics will include: Ppeak , Pplat (Plateau pressure), Cdin (Dynamic Compliance), Cstat (Static Compliance) and DP (Driving pressure). The measurements will be taken in dynamic conditions (Ppeak and Cdin) and by using the maneuver of extending the inspiratory pause to 40% of the length of inspiration, in static conditions, Pplat and Cstat values will be obtained. DP will be calculated according to the formula DP = Pplat - PEEP.

From the hemodynamic measurements, changes in mean arterial pressure (MAP) and heart rate (HR) in the mentioned 6 time points T1 - T6 will be monitored. Arterial blood gas analyzes will be sampled 2 times during the surgical procedure, before the first recruitment maneuver and after the second recruitment maneuver.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years of age
* ASA score ≤ 3 (American Society of Anesthesiologists Physical Status)
* scheduled for laparoscopic cholecystectomy

Exclusion Criteria:

* patients under the age of 18
* pregnant women
* ASA status ˃ 3,
* BMI < 18.5, and ≥ 35 kg/m2
* previous open abdominal surgery
* previous lung surgery
* obstructive and restrictive lung diseases
* neuromuscular diseases
* hemodynamic instability during recruitment maneuver (drop in systolic blood pressure by more than 20% compared to basal values or systolic blood pressure < 90 mmHg)
* bradycardia (drop in heart rate by more than 20% or frequency < 50/min)
* decrease in saturation (SpO2 ≤ 92% for more than 1 minute) during the recruitment maneuver

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Static compliance | 3 hours
  Cstat = VT / (Pplat - PEEP)

SECONDARY OUTCOMES:
Mean arterial pressure | 3 hours
  MAP = (SBP + 2*DBP) / 3
Arterial blood oxygen level | 3 hours
  Partial pressure of oxygen in arterial blood gas analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical center of Vojvodina, Novi Sad, Serbia